CLINICAL TRIAL: NCT00192998
Title: The Serotonergic Transmitter System in Dementia and Affective Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: SERT-AD
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2005-09

CONDITIONS: Mood Disorders; Alzheimer Disease
Keywords: Affective disorder; Alzheimer dementia; healthy controls
MeSH Terms: conditions — Mood Disorders; Alzheimer Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The aim of this project is to examine the serotonergic transmitter system using functional imaging of the brain (positron emission tomography [PET]) to gain knowledge about early pathophysiological changes in Alzheimer's dementia and mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Alzheimer's disease
* Individuals genetically predisposed to affective disorder
* Healthy gender and age matched controls

Exclusion Criteria:

* Contraindications to magnetic resonance imaging (MRI)
* Use of psychoactive drugs
* Past or present affective disorder
* Other systemic diseases that may affect brain function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Vibe G. Frokjaer, MD, Principal Investigator — Neurobiological Research Unit, Copenhagen University Hospital, Denmark
Locations (1):
- Neurobiological Research Unit, Copenhagen, Denmark

REFERENCES:
- See also: homepage for the neurobiological research unit, Copenhagen, Denmark — http://www.nru.dk